CLINICAL TRIAL: NCT01823354
Title: Executive Dysfunction in Restless Legs Syndrome: Determination of Clinical Correlates and Outcome After Therapeutic Management
Brief Title: Executive Dysfunction in Restless Legs Syndrome: Clinical Correlates and Outcome After Therapeutic Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 8964
Record Dates: First submitted 2013-03-22; First posted 2013-04-04 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; Polysomnography; Executive cognition
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients (Other): Polysomnography, Assessment of executive functions, Clinical scales, Medical consultation
  Interventions: Other: Polysomnography; Other: Clinical Scales; Other: Assessment of executive functions; Other: Medical consultation
- Controls (Other): Polysomnography, Assessment of executive functions, Clinical scales Medical consultation
  Interventions: Other: Polysomnography; Other: Clinical Scales; Other: Assessment of executive functions; Other: Medical consultation

INTERVENTIONS:
Other: Polysomnography — Polysomnography involves the collection of the electroencephalogram, electromyogram of, and electro-oculogram to differentiate the various stages of sleep. Determination of different stages and cycles of sleep will be manually by reading the EEG, EMG, EOG over periods of 30 seconds after the standardized criteria of AASM (American Academy of Sleep Medicine). Registration will take place between sleep and 23h 7am.
Other: Clinical Scales — Index of Restless Legs Syndrome Severity, Index of insomnia Severity, Beck's Inventory of Depression, Anxiety Inventory: State-Trait, form Y.
Other: Assessment of executive functions — Verbal fluencies Test GREFEX (Assessment of the spontaneous flexibility), Stroop Test GREFEX (Inhibition of the automatic response Capacity ), Trail Making Test GREFEX (Assessment of flexibility "reactive"), Wisconsin Card Sorting Test(Overall assessment of executive functions), Working memory TAP, Flexibility TAP, Go/no go TAP, Phasic alertness (Assessment of speed information processing).
Other: Medical consultation — open questions

SUMMARY:
Restless leg syndrome (RLS) is a common neurological disorder whose diagnosis is only clinical. The efficacy of dopaminergic agents in improvement of sensorimotor symptoms advance the hypothesis that altered dopaminergic transmission is at the origin of this condition. RLS usually leads to a sleep fragmentation, which induces sometimes severe insomnia most often associated, in clinical practice, to a cognitive complaint (attentional in nature). Executive functions in which dopaminergic transmission is heavily involved refer to a set of complex functions. At least three of them should be considered during their evaluation (ie flexibility, inhibition, and the updating of working memory). These functions are among the targets of the alteration of the quality and quantity of sleep. The few studies that have focused on the study of the integrity of executive functions in RLS have discordant results. The lack of control of key variables in the assessment of executive functioning (ie intellectual performance, depressive symptomatology, generalized slowing in information processing) and the lack of reference in the theoretical approach in executive functions are certainly the two main reasons. Moreover, the question of polysomnographic correlates and the reversibility of these cognitive abnormalities after pharmacological management of RLS remains unanswered today.

The main objective of this study is to compare the executive performance of untreated RLS patients with a group of matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific criteria (patients and controls)

  * Age: 18 to 70 years old
  * Fluency in French (written and oral);
  * intellectual performance within the normal range (f-NART> 84)
  * Subject has signed and returned to the investigator a copy of the signed informed consent; .Affiliated to a social security scheme.
* Specific criteria patients

  * Response to the diagnostic criteria established by the standards of the ICSD-II (2005) and IRLS Study Group (2003) with a severity scale listed at least 21 (score at least severe);
  * MPMS score> 10 / h; .ferritin > 50 ng/ml.

Exclusion Criteria:

* Exclusion criteria (patients and controls)

  * Taking any psychotropic medication within 15 days prior to polysomnography (except for patients on dopamine agonist reassessed at 6 months follow-up);
  * Pregnant and lactating women;
  * Pneumologic affection
  * Night shift;
  * Apnea-hypopnea index > 15; .Major subjects protected by the law, under guardianship.
* Exclusion criteria (controls)

  * Neurological or psychiatric current and/or past;
  * MPMS score> 10 / h; .Subject currently participating in another clinical research project prohibiting joint participation in another biomedical research, or who are in a period of exclusion or who have already received the maximum legal compensation for stresses in the year.
* Exclusion criteria (patients)

  * Presence of other neurological conditions present and / or a psychiatric disorder (other than a mood disorder and / or anxiety); .RLS patients previously treated with a dopamine agonist who has not stopped treatment at least 15 days before the start of the study.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2012-11-26 (Actual); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Verbal fluency test between untreated RLS patients and control subjects | Day 0
  Number of correct words (without repetitions and intrusions) provided by the subject in each condition.

SECONDARY OUTCOMES:
Change of the Clinical Scales at day 180 (composite criteria) | Day 0 and day180
  * Index of Restless Legs Syndrome Severity
  * Index of insomnia Severity
  * Beck's Inventory of Depression
  * Anxiety Inventory: State-Trait, form Y
Change of the sleep fragmentation at day 180 (composite criteria) | Day 0 and Day 180
  The severity of sleep fragmentation is determined by these parameters:
  * Total time asleep in minutes.
  * Percentage of sleep efficiency.
  * Ensure intra-sleep.
  * Index of arousals / hour of sleep.
  * Index of periodic movements per hour of sleep associated with arousal
  * Index of arousal.
Assessment of executive functions (composite criteria) | Day 180
  * Trail Making Test GREFEX
  * Sroop Test GREFEX
  * Wisconsin Card Sorting Test
  * Phasic alertness TAP
  * Working memory TAP
  * Flexibility TAP
  * Go / no go TAP
  * Score of Reached Executive Severity
Change of the Verbal fluency test after dopamin agonist treatment in RLS patients | Day 0 and Day 180
  Number of correct words (without repetitions and intrusions) provided by the subject in each condition.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Dauvilliers, PU, PH, Principal Investigator — UH Montpellier
Locations (2):
- France (2):
  - UH Montpellier, Montpellier
  - UH Nîmes, Nîmes